CLINICAL TRIAL: NCT00194948
Title: Patient Preference in Primary Care Depression Treatment
Brief Title: Treatment Choices for Improving Adherence and Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH069784 (NIH); K23MH069784 (NIH); DSIR 8K-RTSE
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Interpersonal Psychotherapy

INTERVENTIONS:
Drug: escitalopram
Behavioral: interpersonal psychotherapy

SUMMARY:
This study will determine the effectiveness of offering primary care patients their preferred treatment versus one that is less desirable in improving treatment adherence and outcome.

DETAILED DESCRIPTION:
This study investigates whether offering primary care patients treatment that is congruent with their preferred first choice improves adherence and outcomes, in comparison to offering treatment that is not congruent with their preferred first choice. All subjects are offered a treatment with demonstrated efficacy, namely either the antidepressant medication escitalopram or Interpersonal Psychotherapy for 5 months. We hypothesize that patients who receive congruent treatment will be more likely to initiate treatment, adhere to treatment, and achieve depression remission.

ELIGIBILITY:
Inclusion Criteria:

* age 21-99
* English-speaking
* DSM-IV criteria for major depression

Exclusion Criteria:

* unable to give informed consent
* MMSE<24
* DSM-IV diagnosis of bipolar disorder, psychotic disorder, current alcohol or substance abuse
* active suicide ideation
* aphasia
* acute or severe medical illness
* currently receiving either antidepressant medication or psychotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
treatment initiation
treatment adherence

SECONDARY OUTCOMES:
depressive symptomatology

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Raue, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Cornell Internal Medicine Associates, New York, New York
  - Weill Medical College of Cornell University, White Plains, New York